CLINICAL TRIAL: NCT05634772
Title: Dormia Basket Versus Extraction Ballon in Proximally Migrated Biliary Stents:A Randomized Controlled Clinical Trial
Brief Title: Dormia Basket Versus Extraction Ballon in Proximally Migrated Biliary Stents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohammed Hussien Ahmed, Clinical professor, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kafrelsheikh U , medicine
Record Dates: First submitted 2022-11-09; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Biliary Obstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the efficacy of dormia basket in management of proximal stent migration (Active Comparator)
  Interventions: Device: dormia basket
- the efficacy of extraction biliary balloon in management of proximal stent migration (Active Comparator)
  Interventions: Device: Extraction biliary ballon

INTERVENTIONS:
Device: dormia basket — Use of dormia basket in management of proximal stent migration
  Arms: the efficacy of dormia basket in management of proximal stent migration
Device: Extraction biliary ballon — Use of extraction biliary balloon in management of proximal stent migration
  Arms: the efficacy of extraction biliary balloon in management of proximal stent migration

SUMMARY:
Dormia basket versus extraction ballon in proximally migrated biliary stents:A randomized controlled clinical trial

DETAILED DESCRIPTION:
Dormia basket versus extraction ballon in proximally migrated biliary stents:A randomized controlled clinical trial The study aims to evaluate the efficacy of dormia basket versus extraction biliary balloon in management of proximal stent migration

ELIGIBILITY:
Inclusion Criteria:

1. Adults
2. both gender
3. Patients with biliary stenting following ERCP and who had signs of biliary obstruction.

Exclusion Criteria:

ERCP without stent insertion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
To compare between dormia basket and extraction ballon in management of proximally migrated biliary stents regarding operative time (min) | 4 weeks
  Operative time was measured by minutes

OTHER OUTCOMES:
To compare between dormia basket and extraction ballon regarding occurrence of re- obstruction | 4 weeks
  Re-obstruction was measured by serum bilirubin level

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Hussien Ahmed, Kafr ash Shaykh, Egypt